CLINICAL TRIAL: NCT01883440
Title: A Placebo Controlled Study With a Nasal Spray Containing Glucose Oxidase, Aiming to Induce a Faster Recovery From an Episode of Common Cold
Brief Title: Glucose Oxidase as Treatment Against Common Cold
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Krister Tano (Other)
Responsible Party: Sponsor-Investigator, Krister Tano, MD, PhD, Umeå University
Organization: Umeå University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GOcoldSY2013
Record Dates: First submitted 2013-04-23; First posted 2013-06-21 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2015-12

CONDITIONS: Common Cold
Keywords: Duration
MeSH Terms: conditions — Common Cold | interventions — Glucose Oxidase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline+glucose (Placebo Comparator): A nasal spray with isotone saline + 5% glucose in a bag-on-valve nasal spray device. The spray will be administered with one puff in each nostril 5 times day one and thereafter trice daily for a total treatment time of one week
  Interventions: Drug: Saline+glucose
- Glucose oxidase + glucose (Active Comparator): A nasal spray (bag-on-valve device) with 200U/ml glucose oxidase + 5% glucose in isotone saline. One puff in each nostril 5 times daily day one and 3 times daily thereafter. A total treatment time of one week.
  Interventions: Drug: Glucose oxidase + glucose

INTERVENTIONS:
Drug: Glucose oxidase + glucose — Isotone saline + 200U/ml of glucose oxidase + 5% of glucose in a bag on valve nasal spray device
  Arms: Glucose oxidase + glucose
Drug: Saline+glucose — Placebo arm
  Arms: Saline+glucose

SUMMARY:
Glucose oxidase is a hydrogen peroxide producing enzyme, which also is present in honey. Human rhinoviruses are sensitive to the action of hydrogen peroxide, which is documented in laboratory studies.

In the present study we aim to investigate if a nasal spray with glucose oxidase could treat a common cold, when the treatment is started even after the onset of the symptoms. The study is randomized and placebo controlled.

DETAILED DESCRIPTION:
Persons that are convinced of that they have caught an episode of common cold can be included into the study within 24 hours after the onset of symptoms.

Before they start the treatment with the nasal spray they perform a viral sample from the nose and also fill in the WURSS-21 protocol. After this the persons spray with glucose oxidase+glucose/only saline+glucose 5 times the first day and thereafter 3 times daily for a total treatment of one week. Every day the included persons fill in the WURSS-21 protocol.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of a common cold within the last 24 hours

Exclusion Criteria:

* Use of a nasal steroid due to allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Toolanen, MD, Study Chair — Norrbottens Läns Landsting
Locations (1):
- Öronmottagningen, Södra Sunderbyn, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline+Glucose: A nasal spray with isotone saline + 5% glucose in a bag-on-valve nasal spray device. The spray will be administered with one puff in each nostril 5 times day one and thereafter trice daily for a total treatment time of one week
  saline+glucose: Isotone saline+5%glucose in a bag-on-valve nasal spray device
Period: Overall Study
Arm/Group | Saline+Glucose | Glucose Oxidase + Glucose
Started | 45 | 45
Completed | 42 | 45
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: All persons that completed the 7 Days of treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline+Glucose | Glucose Oxidase + Glucose | Total
Number analyzed (Participants) | 42 | 45 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 45 | 87
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 44 [18 to 63] | 41 [21 to 61] | 42 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 35 | 68
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  Sweden | 42 | 45 | 87

OUTCOME MEASURES:

1. Primary Outcome: Sum of All Symptoms in Viruspositive Persons
Description: Symptoms of a common cold, recorded in a home protocol, "Wisconsin Upper Respiratory Symptom Score 21 (WURSS21)" daily for 7 days was used as the evaluation method of the treatment. WURSS-21 is a validated protocol for assessing symptoms of a common cold. We used this protocol at start, before the persons in the study started their treatment and thereafter every day for the next 7 days. WURSS 21 consists of 21 questions (last question is not valid) regarding different symptoms as: running nose, sore throat, cough, blocked nose, etc. Every such question is graded from 0-7, 0 is defined as no such symptom and the number 7 means the worst possible symptom. The outcome measure is predominantly calculated as "the sum of all symptoms" in the WURSS-21 protocol, which means that the value from each of the 20 questions (min=0, max=140) is summarized every day for each of the participants, which gives a mean value for both groups every day.
Time Frame: One week
Population: The persons analyzed were those that had a positive viral sampling with Parainfluenza, Corona or Rhinoviruses, that is: the viruses that most often causes common cold and also would be accessible for treatment with a nasal spray.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Saline+Glucose | Glucose Oxidase + Glucose
Number analyzed (Participants) | 14 | 13
units on a scale
  Start value | 52 [8 to 63] | 52 [18 to 92]
  Value day 1 | 54 [8 to 84] | 56 [14 to 81]
  Value day 2 | 58 [13 to 95] | 53 [8 to 108]
  Value day 3 | 52.5 [7 to 80] | 38 [2 to 106]
  Value day 4 | 48 [2 to 83] | 31 [0 to 87]
  Value day 5 | 39 [0 to 99] | 26 [0 to 71]
  Value day 6 | 36 [0 to 96] | 18 [0 to 77]
  Value day 7 | 29 [0 to 61] | 14 [0 to 72]
Statistical Analysis 1: Comparison: Saline+Glucose vs Glucose Oxidase + Glucose; Test type: Superiority or Other; p < 0.037, Mixed Models Analysis; Linear mixed model

2. Primary Outcome: Sum of All Symptoms of All Persons That Fullfilled the Study
Description: as for outcome 1
Time Frame: 7 days
Population: All of the persons that fullfilled the study
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Saline+Glucose | Glucose Oxidase + Glucose
Number analyzed (Participants) | 42 | 45
units on a scale
  Start | 42 [4 to 81] | 42 [4 to 99]
  Day 1 | 44 [5 to 84] | 42 [6 to 104]
  Day 2 | 45 [0 to 95] | 39 [0 to 121]
  Day 3 | 40 [0 to 84] | 34 [0 to 123]
  Day 4 | 33 [0 to 83] | 31 [0 to 118]
  Day 5 | 27 [0 to 99] | 27 [0 to 74]
  Day 6 | 21 [0 to 96] | 23 [0 to 78]
  Day 7 | 17 [0 to 61] | 19 [0 to 78]
Statistical Analysis 1: Comparison: Saline+Glucose vs Glucose Oxidase + Glucose; In the material when all were included, there were a lot of persons with few symptoms in both Groups, which means that a larger study would be needed in order to detect significant differences; Test type: Superiority or Other; p = 0.381, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Saline+Glucose | Glucose Oxidase + Glucose
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

LIMITATIONS AND CAVEATS:
Viral samplings were made in order to exclude persons with no viral infection and persons with influenza. Most common Colds are due to Rhinoviruses, Parainfluenza and Coronaviruses. These persons were included in the Groups with significant findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No